## **Statistical Analysis plan**

The collected data was tabulated and analyzed using Statistical Package for Social Science (SPSS 15.0 for windows; SPSS Inc, Chicago, IL, 2001). First; the normality of distribution of parameters was evaluated by One-Sample Kolmogrovo-smirnov test. Data were expressed as mean and standard deviation (SD). One-Way ANOVA test was used for comparison between more than two study group means. Pairwise multiple comparisons to test the difference between each pair of means was performed using Tukey HSD test, and yield a matrix where different asterisks indicate significantly different group means. Paired t test was used to compare changes within same group. For all tests, P <0.05 was considered significant.